CLINICAL TRIAL: NCT03562039
Title: Clinical and Radiographic Evaluation of Intra Bony Defects Following Complete Versus Incomplete Removal of Granulation Tissue in Modified Minimally Invasive Surgical Technique (M-MIST). A Randomized Controlled Clinical Trial.
Brief Title: Evaluation of Healing of Intra-bony Defects in Modified Minimal Invasive Surgical Technique
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ahmed Ibrahim, principle investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 125896
Record Dates: First submitted 2018-05-22; First posted 2018-06-19 (Actual); Last update posted 2024-03-05 (Actual); Status verified 2024-03

CONDITIONS: Periodontal Regeneration, Clinical and Radiographic Results, Modified Minimal Invasive Surgery

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- M-MIST (group A) (Experimental): M-MIST(incomplete granulation tissue removal)
  Interventions: Procedure: M-MIST
- M-MIST (group B) (Active Comparator): conventional M-MIST.
  Interventions: Procedure: M-MIST

INTERVENTIONS:
Procedure: M-MIST — minimal invasive surgical technique without thorough removal of granulation tissue

SUMMARY:
This study is aiming to compare the clinical and radiographic outcomes after complete versus incomplete removal of granulation tissue during modified minimally invasive surgical technique for management of periodontal intrabony defects in patients with chronic periodontitis.

DETAILED DESCRIPTION:
Periodontal surgery has been expanding in the world of dentistry throughout the past years, as new techniques are emerging to treat the different and complex periodontal disorders. Surgical procedures in dentistry have undergone major changes to minimize invasiveness. In addition, novel instruments and materials have been made to suit the evolution of the surgical procedures (Cortellini. 2012).

Teeth with deep pockets associated with deep intra-bony defects are a clinical challenge for periodontists, where periodontal regeneration has been proven to be effective in managing the treatment of one-, two-, and three-wall intra-bony defects (Needleman and Tucker 2012;Needleman. 2015).

Harrel and Rees (1995) were the first to introduce the term minimally invasive surgery (MIS). MIS is used to describe the use of smaller and more precise surgical procedures that are possible by using of magnifying instruments, such as operating microscopes and microsurgical instruments and materials (Cortellini. 2012).

The rationale for the development of minimally invasive surgical technique (MIST) includes: reduction of trauma during the surgery, increase in flap and wound stability, improvement of wound primary closure, reduction of surgical time, and minimization of intra-operative and post-operative patient discomfort (Cortellini. 2007).

With the use of MIST, Cortellini and Tonneti (2009) confirmed blood clot protection with the aspects of wound and blood clot stability and primary wound closure.

An enhancement of MIST, the modified minimally invasive surgical technique (M-MIST), has been introduced by Cortellini in 2009 to further reduce the surgical invasiveness, with three major objectives in mind: (1) minimize the interdental tissue tendency to collapse providing space provision for regeneration, (2) enhance the wound/soft tissue stability and (3) reduce patient morbidity.

Some authors evaluated the use of various regenerative material in MIST and M-MIST e.g. Enamel matrix derivative (Cortellini 2007) PDGF-bb (Cosyn et al. 2012) and collagen enriched bovine derived xeno-graft (Mishra et al., 2013). Cortellini (2011) also, noted that the use of regenerative material is not necessary with M-MIST.

Hung et al, (2012) reported that granulation tissue could contain progenitor stem cells which are very important components needed for periodontal tissue regeneration.

Moreover, Park et al. (2011) assumed that the inflamed granulation tissue could be used to regenerate lost tissues in the same individual in other defective sites according to its regenerative potential.

All the previous data raised an important question about the necessity to remove granulation tissues in periodontal regenerative techniques: Is complete removal of granulation tissue in M-MIST is mandate for treating isolated intra-bony defects for better healing?

ELIGIBILITY:
Inclusion Criteria:

* - systemically healthy patients
* Age range from 25 - 55.
* Patients with moderate to advanced chronic periodontitis with pockets ≥ 5 mm 6-8 weeks after phase I (non-surgical) therapy.
* Vertical 2 or 3 walls Intra-bony defects.
* Perform and maintain good oral hygiene.
* Able to come for the follow up appointment's needed

Exclusion Criteria:

* - Smokers.
* Pregnant patients.
* patients with poor oral hygiene.
* Multirooted teeth with furcation involvement.

Ages: 25 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2018-04-15 (Actual); Primary Completion 2021-03-30 (Actual); Study Completion 2021-04-03 (Actual)

PRIMARY OUTCOMES:
changes in clinical attachment level | at baseline then 6, 9 and 12 months
  It is the distance from the cement-enamel junction to the depth of the pocket.

SECONDARY OUTCOMES:
changes in pocket probing depth | at baseline then at 6, 9 and 12 months
  distance from the depth of the pocket to the gingival margin
changes in gingival recession | at baseline then at 6, 9 and 12 months
  distance of the exposed root surface from the cemento-enamel junction to the gingival margin
amount of bone fill | at baseline then at 6, 9 and 12 months
  difference in bone fill in standardized periapical radiograogh
patient pain and discomfort | at day of the surgery then at 1 , 3 and 7 days post-surgery
  by giving the patient a questionnaire to fill
patient satisfaction | 12 months post-surgery
  by giving the patient a questionnaire to fill

CONTACTS AND LOCATIONS:
Overall Officials: Hani Nahass, Ass.prof., Study Director — Cairo University
Locations (2):
- Egypt (2):
  - Cairo University, Cairo, Manyal
  - Cairo University, Giza

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol

REFERENCES:
- [Background] Cortellini P, Tonetti MS. Improved wound stability with a modified minimally invasive surgical technique in the regenerative treatment of isolated interdental intrabony defects. J Clin Periodontol. 2009 Feb;36(2):157-63. doi: 10.1111/j.1600-051X.2008.01352.x. PMID 19207892
- [Background] Ainamo J, Bay I. Problems and proposals for recording gingivitis and plaque. Int Dent J. 1975 Dec;25(4):229-35. PMID 1058834
- [Background] Fickl S, Thalmair T, Kebschull M, Bohm S, Wachtel H. Microsurgical access flap in conjunction with enamel matrix derivative for the treatment of intra-bony defects: a controlled clinical trial. J Clin Periodontol. 2009 Sep;36(9):784-90. doi: 10.1111/j.1600-051X.2009.01451.x. Epub 2009 Jul 14. PMID 19614721
- [Background] Ramfjord SP. The Periodontal Disease Index (PDI). J Periodontol. 1967 Nov-Dec;38(6):Suppl:602-10. doi: 10.1902/jop.1967.38.6.602. No abstract available. PMID 5237683
- [Background] Bajaj P, Agarwal E, Rao NS, Naik SB, Pradeep AR, Kalra N, Priyanka N, Kumari M. Autologous Platelet-Rich Fibrin in the Treatment of 3-Wall Intrabony Defects in Aggressive Periodontitis: A Randomized Controlled Clinical Trial. J Periodontol. 2017 Nov;88(11):1186-1191. doi: 10.1902/jop.2017.120661. Epub 2017 Aug 18. PMID 28820320
- [Background] Patel GK, Gaekwad SS, Gujjari SK, S C VK. Platelet-Rich Fibrin in Regeneration of Intrabony Defects: A Randomized Controlled Trial. J Periodontol. 2017 Nov;88(11):1192-1199. doi: 10.1902/jop.2017.130710. Epub 2017 Aug 18. PMID 28820322
- [Background] Harrel SK. 1999. "A Minimally Invasive Surgical Approach for Periodontal Regeneration: Surgical Technique and Observations. J Periodontol 70: 1547-1557." Hung, Tzu-yuan, Hsiang-chun Lin, and Ying-jen Chan. 2012. "Isolating Stromal Stem Cells from Periodontal Granulation Tissues," 1171-80. doi:10.1007/s00784-011-0600-5. J-c, Park, Kim J-m, Jung I-h, Kim Jc, Choi S-h, Cho K-s, Kim C-s Isolation, and Chang-sung Kim. 2011. "Isolation and Characterization of Human Periodontal Ligament ( PDL ) Stem Cells ( PDLSCs ) from the Inflamed PDL Tissue : In Vitro and in Vivo Evaluations" 18: 721-31. doi:10.1111/j.1600-051X.2011.01716.x. Lindhe and Nyman, periodontology Clinical. 1985. "Scaling and Granulation Tissue Removal in Periodontal Therapy *," no. 1983: 374-88. Needleman, I. 2015. "Clinical Concepts for Regenerative Therapy in Intrabony Defects" 68: 282-307.
- [Result] Cortellini P, Tonetti MS. Clinical and radiographic outcomes of the modified minimally invasive surgical technique with and without regenerative materials: a randomized-controlled trial in intra-bony defects. J Clin Periodontol. 2011 Apr;38(4):365-73. doi: 10.1111/j.1600-051X.2011.01705.x. Epub 2011 Feb 8. PMID 21303402